CLINICAL TRIAL: NCT06648837
Title: Continuous Blood Donation for the Development of the Microvisk PT/INR
Brief Title: Microvisk Continuous Blood Donation Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Microvisk Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PJP-R-0005
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Embolism (Diagnosis); Deep Vein Thrombosis; Atrial Fibrillation (AF)
Keywords: PT; INR; PT/INR; Warfarin; Vitamin K agonist; POC testing
MeSH Terms: conditions — Pulmonary Embolism; Disease; Venous Thrombosis; Atrial Fibrillation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Warfarin patients (Experimental): Single Arm - blood collection by venepuncture in patients undergoing Warfarin Therapy
  Interventions: Procedure: Venepuncture; Other: Collection of relevant information

INTERVENTIONS:
Procedure: Venepuncture — Venepuncture to collect blood samples from Patients undergoing Warfarin Therapy, additional tubes of blood drawn during normal clinical vist.
Other: Collection of relevant information — Collect relevant information to ensure potential participant meets all inclusion/exclusion criteria.

SUMMARY:
Microvisk Technologies Ltd designs and develops test systems for monitoring the effectiveness of Warfarin and Warfarin-like medications.

Warfarin and Warfarin-like medications are used to reduce the risk of stroke in people with an irregular heart rhythm (Atrial Fibrillation) or with mechanical heart valve replacements, as well as reducing the risk of recurrent Venous Thromboembolism.

Warfarin dosing needs to be individualized. In order to correctly dose an individual in order to optimize the effectiveness of warfarin, and minimize the risk of bleeding, close monitoring of the degree of anticoagulation is required through regular blood testing. This test is known as PT/INR (Prothrombin Time/International Normalised Ratio). Simply, it is the measure of the amount of time (in seconds) it takes for your blood to clot.

Microvisk Technologies Ltd are developing new anticoagulant test strips for patients on warfarin or warfarin like medications. The blood collected as part of this study will be tested upon Microvisk's second generation Prothrombin/International Normalized Ratio (PT/INR) Test System. The donated blood will be used on ongoing development, validation, verification, and calibration projects. This study is being performed in partnership with the Oxford University Hospital (OUH) and Local Clinical Research Networks (LCRN) Thames Valley Core team, part of National Institute for Health and Care Research (NIHR).

DETAILED DESCRIPTION:
The number of patients receiving anticoagulation therapy with warfarin and other vitamin K antagonists has been rising in recent years. Increasing life expectancy is increasing the proportion of the population having conditions such as Atrial Fibrillation and venous thrombosis, where primary and secondary prevention of thromboembolic complications are best achieved with anticoagulation.

Unpredictable pharmacokinetics, widespread interactions with drugs and food and the narrow therapeutic window make closely monitoring Vitamin K antagonists a necessity. Portable point of care (POC) coagulometers which measure PT from capillary whole blood and provide an INR reading within a few minutes are already widely available throughout North American and Europe. They give comparable results when compared to laboratory based systems are popular with patients and significantly shorten the duration of clinics. In addition, the United Kingdom Department of Health has been encouraging the use of anticoagulation services in Primary Care Trusts the aim being to provide INR monitoring in community clinics and General Practice surgeries relieving pressure on hospital services and reducing inconvenience for patients.

Although coagulometers are now commercially available the Microvisk INR Testing System has been designed to have advantages, particularly in terms of test robustness, user comfort, ease of use and reduction of user error. The present trial has been designed to develop the second generation Microvisk INR Test System; blood samples will also be used to optimise manufacturing processes and verify the quality of Test Strip Lots.

ELIGIBILITY:
Inclusion Criteria:

* Currently undergoing Warfarin therapy.
* Over 18 years old

Exclusion Criteria:

A participant is not eligible for participation if ANY of the following criteria are met:

* Participant is <18 years of age
* Participant is unable to give consent
* Participant has been treated with Unfractionated Heparin, or Low Molecular Weight Heparin, within the last 7 days
* Participant has, or is suspected of having, Anti-Phospholipid Syndrome (APS)
* Participant is pregnant, or has been in the past 12 months
* Participant is known to have HIV/AIDS, is a carrier of Hepatitis A, B or C, has had tuberculosis or a tropical disease
* Participant is suspected of intravenous drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2025-01-13 (Estimated); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Ongoing development of Microvisk Technologies PT/INR products | 5 years
  The Primary Outcome will be measured in terms of differences in International Normalised Ratio when the Generation 2 CoagMax system is tested against the lab benchtop analyser using the blood samples from the same donors.
  Those differences will be reported in terms of accuracy, precision and sensitivity to interferents.

SECONDARY OUTCOMES:
The Secondary Outcome will be measured in terms of differences in International Normalised Ratio when the Generation 2 system is tested against the International Standard Method using the blood samples from the same donors. | 5 years
  A master batch of test strips will be calibrated against an International Reference Preparation (rTF/09) thromboplastin. The accuracy of the master batch will be verified using patient samples.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shapiro, Principal Investigator — Oxford Haemophilia and Thrombosis Centre Oxford University Hospital NHS Foundation Trust
Locations (1):
- Oxford Haemophilia and Thrombosis Centre, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No